CLINICAL TRIAL: NCT05231603
Title: Randomized, Double Blind, Placebo Controlled Clinical Trial of Ivermectin For Post Exposure Prophylaxis For COVID-19 Infection Among Close Contacts
Brief Title: Ivermectin for Post Exposure Prophylaxis of Covid-19
Acronym: I-CPEP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor response
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Hovid Berhad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NMRR-21-1371-60569
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Ivermectin; Post exposure; Prophylaxis
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: This is a randomized, double blind, placebo controlled clinical trial evaluating the effect of Ivermectin for post exposure prophylaxis among close contacts of COVID-19 positive case patient as an index case.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group: (Active Comparator): Ivermectin 0.4 mg/kg/day (maximum 24 mg)
  Interventions: Drug: Ivermectin
- Control group (Placebo Comparator): Placebo-inactive substance
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin — 0.4 mg/kg/day-maximum dose is 24 mg.
  Arms: Treatment group:
Other: Placebo — Similar to drug in term of tablets
  Arms: Control group

SUMMARY:
Post exposure prophylaxis of healthy contacts is among the measures used for outbreak control of several infectious diseases (e.g., pandemic influenza). No agent is known to be effective in preventing COVID-19, but Ivermectin is one of the drugs that have shown antiviral activity against SARS-CoV-2 in the laboratory. This study aims to evaluate the effect of post exposure prophylaxis with Ivermectin after exposure to COVID-19 among the asymptomatic close contacts.

DETAILED DESCRIPTION:
Primary Objective:

To assess the efficacy of Ivermectin as post exposure prophylaxis in asymptomatic adults (≥18 years of age) who had close-contact exposure to a confirmed case of COVID-19 patient

Secondary Objectives:

1. To compare the viral load (using CT value reading) among close contacts who become positive COVID-19 during follow up period between the Ivermectin and placebo group
2. To assess the adverse effects of Ivermectin within 7 days after each dose

Study Population and Sampel Size Asymptomatic adults (≥18 years of age) who had recent history (less than 5 days) of close contact exposure to a confirmed COVID-19 positive patient as per the definition by CDC.

In this study, the study teams decide to recruit 150 subjects per group, a total of 300 subjects; 30 subjects in each site (15 Ivermectins, 15 placebos)

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic individuals exposed to a confirmed positive COVID-19 case within 5 days from the study recruitment day (include household, workplace and social close contact)
2. Aged ≥18 years; male or female
3. No fever with temperature less than 37.5ºC
4. RTK Ag for COVID-19 is negative on the recruitment day.
5. For subject who had received COVID-19 vaccination:

   * Any primary series vaccine (eg: Pfizer, Sinovac, AstraZeneca etc) : past 90 days after the second dose
   * Any booster vaccine: past 90 days after the booster dose
6. In women of childbearing potential (18-55 years old), negative pregnancy test and agree to use any contraceptive method up to 7 days after the second dose of IP administration
7. Have access to video and phone call
8. Willing to take 2 doses of study medication (2 days apart between Dose 1 and Dose 2)
9. Willing to comply with all study procedures
10. Able to provide written informed consent

Exclusion Criteria:

1. Unable to take drugs by mouth
2. History of positive confirmed COVID-19 infection within past 3 months
3. Involved in any COVID-19 vaccine clinical trial
4. Patients with suspected concomitant bacterial, fungal infections, concurrent congestive heart failure prior to initiation of study drug
5. Known case of liver disease (any severity)
6. Alcohol intake more than recommended (2 drinks or more in a day for men and 1 drink or more in a day for women)
7. Mal-absorption syndrome or other clinically significant gastrointestinal disease that may affect absorption of the study drug (non-correctable vomiting, diarrhea, ulcerative colitis, and others).
8. Pregnant or nursing/breastfeeding women or women planning for pregnancy.
9. Female patients who cannot consent to contraceptive use (any method) from the start of IP administration to 7 days after the second dose of IP administration
10. Male patients whose partner cannot agree to use the contraception method as in 9)
11. Patients with a history of gout or on treatment for gout or hyperuricemia
12. Patients receiving immunosuppressant
13. Patients who have previously received Ivermectin.
14. Patients who are not able to provide written consent.
15. Other patients judged ineligible by the principal investigator or sub-investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Female
Enrollment: 50 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Number of Covid-19 cases | 8 weeks
  Comparison of the number of confirmed COVID-19 cases among the close contacts after exposure to a confirmed case of COVID-19 patient in Ivermectin and placebo group

SECONDARY OUTCOMES:
CT value in Covid-19 | 14 days
  Comparison of the CT value between Ivermectin and placebo group

OTHER OUTCOMES:
Adverse effects of Ivermectin | 14 days
  To assess the adverse effects of Ivermectin within 7 days after each dose

CONTACTS AND LOCATIONS:
Locations (10):
- Malaysia (10):
  - KK Bandar Sg Petani, Sungai Petani, Kedah
  - KK Bagan Serai, Bagan Serai, Perak
  - KK Greentown, Ipoh, Perak
  - KK Karai, Kuala Kangsar, Perak
  - KK Ayer Tawar, Sitiawan, Perak
  - KK Tanjung Malim, Slim River, Perak
  - KK Simpang, Taiping, Perak
  - KK Tapah, Tapah, Perak
  - KK Kangar, Kangar, Perlis
  - KK Seberang Jaya, Butterworth, Pulau Pinang

IPD SHARING:
Plan to Share IPD: No